CLINICAL TRIAL: NCT07030569
Title: RADIomics to Predict HER2 Status And T-DXd Efficacy in Metastatic Breast Cancer: the RADIOSPHER2 Study
Acronym: RADIOSPHER2
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: INT34/24
Record Dates: First submitted 2025-01-07; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-01

CONDITIONS: Radiomic; Radiomics; Breast Cancer Metastatic; Breast Cancer Stage IV; Breast Carcinoma; Breast Neoplasms; Breast Cancer; Breast Cancer With Bone Metastasis; Breast Cancer With Metastatic Bone Disease; Trastuzumab; HER2; HER2 + Breast Cancer; HER2 Positive Breast Carcinoma; HER2-positive Breast Cancer; Her2/Neu Positive Advanced Solid Tumors; HER2/Neu-positive Breast Cancer
Keywords: Radiomics; HER2 expression; Trastuzumab Deruxtecan; Pathomics; HER2 heterogeneity
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival Formalin-Fixed Paraffin-Embedded tumor blocks for transciptomic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Metastatic breast cancer patients underwent tumor biopsy in a metastatic site: A cohort of patients with metastatic breast cancer underwent a liver, lung, pleural or bone biopsy in the metastatic setting at INT with available imaging (CT scan and/or PET-FdG scan), performed from 01Jan2005 to 01Jan2024. A subgroup of this cohort is treated with Trastuzumab Deruxtecan.
  Interventions: Drug: Trastuzumab deruxtecan (DS-8201a)

INTERVENTIONS:
Drug: Trastuzumab deruxtecan (DS-8201a) — A subgroup of the study cohort treated with Trastuzumab Deruxtecan in the metastatic setting

SUMMARY:
RADIOSPHER2 study is a monocentric, retrospective, observational study aiming at identifying a radiomics signature able to predict HER2 expression (0 vs low vs overexpression) and trastuzumab deruxtecan efficacy in metastatic breast cancer patients. The study also encompasses translational analyses and inter-modal correlations in order to provide novel insights about HER2 spatial and temporal heterogeneity, at the macroscopic and microscopic levels.

DETAILED DESCRIPTION:
The primary objective of the study is the identification of a radiomic signature ("radiobiopsy") from several features extracted from radiological images to predict the HER2 status on different specific metastatic sites of metastatic breast cancer patients. Accordingly to the study rationale, it will chosen to analyse images from those metastatic sites usually difficulty to approach with biopsy, such as lung, liver, pleural and bone lesions.

The "radiobiopsy" model will be applied to retrospectively calculate HER2 status from the baseline scan of HER2+ or HER2-low mBC patients underwent any-line trastuzumab deruxtecan (T-DXd) treatment for metastatic disease. The T-DXd PFS of patients assigned to the three cohorts (HER2-0, HER2-low or HER2-overexpressed) based on "radiobiopsy" model will be then calculated and differences among groups will be tested with Cox regression analysis. Clinical characteristics (e.g., number of therapy line for metastatic disease, HR status, HER2 IHC expression) of the same cohort will be extracted from clinical health records, in order to build a multivariate Cox regression model.

To assess the HER2 spatial heterogeneity at intra-tumor microscopic level, pathology slides derived from biopsies of patients enrolled to build the "radiobiopsy" model will be also reviewed from pathologists for HER2 heterogeneity evaluation and digitalized for pathomics analyses. The HER2 heterogeneity will be evaluated by pathologist based on IHC expression and distribution. In order to evaluate if radiomic features can predict HER2 heterogeneity at intra-tumor macroscopic level, a different radiomic model will be developed for this purpose, using the HER2 heterogeneity score assigned by pathologist in the previous task as outcome.

In addition, in order to confirm and quantify inter-lesion HER2 spatial heterogeneity, the features included in the discovered "radiobiopsy" signature will be extracted and the HER2 status calculated for the other metastatic lesions. A correlation analysis between HER2 status assignment from different lesions of the same patients will be performed to quantify the prevalence of HER2 variability among lesions in the cohort. In order to clarify if HER2 heterogeneity at microscopic level is associated with inter-lesion heterogeneity, a single-patient correlations between the heterogeneity pathomic score and the inter-lesion radiomic heterogeneity will be performed.

To have insight into the features included into the "radiobiopsy" model, transcriptomics analysis will be conducted through bulk-RNA sequencing from available tumor FFPE specimens of lung, pleural and liver biopsies. The differential expression of several genes and transcriptomic signatures with known prognostic/predictive relevance, such as immune and metabolic genes and signatures, will be assessed among samples with differently expressed features included in the model. It will allow to dissect tumor biology by finding the biological counterpart of agnostic radiomics features that would remain otherwise unexplained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic breast cancer underwent a liver, lung, pleural or bone biopsy in the metastatic setting, performed from 01Jan2005 to 01Jan2024.

Exclusion Criteria:

* Not available imaging (CT scan and/or PET-FdG scan) in the three months before the biopsy or before the last previous treatment interruption;
* Unknown HER2 status;
* Node, soft tissue or other visceral as biopsy site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of the study will consists with a cohort of patients with metastatic breast cancer underwent a liver, lung, pleural or bone biopsy in the metastatic setting at the Sponsor Institution with available imaging (CT scan and/or PET-FdG scan), performed from 01Jan2005 to 01Jan2024.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
HER2 protein expression | Time of the metastatic biopsy (through study completion, an average of 1 year)
  To identify a radiomic signature ("radiobiopsy") able to predict the HER2 status on a specific metastasic site of mBC patients based on radiologic images (CT scan, PET-FdG)
Progression-Free Survival | From treatment start to disease progression or death (through study completion, up to 5 years)
  To test the accuracy of "radiobiopsy" in predicting PFS in a cohort of metastatic breast cancer patients treated with trastuzumab deruxtecan.

SECONDARY OUTCOMES:
HER2 intratumoral heterogeneity | Time of the metastatic biopsy (through study completion, an average of 1 year)
  To identify a pathomic-based model able to predict intratumoral HER2 heterogeneity on pathology slides of HER2-positive and HER2-low mBC patients
HER2 interlesional heterogeneity | Time of the metastatic biopsy (through study completion, an average of 1 year)
  To test the concordance between intratumoral and inter-lesional HER2 heterogeneity in HER2-positive and HER2-low mBC patients.
Radiomics agnostic features | Time of the imaging next to the metastatic biopsy (through study completion, an average of 1 year)
  To correlate the features included in the radiomic model with the transcriptomics data obtain from bulk-RNAseq from biopsies, in order to explain agnostic features discovered with radiomics.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT07030569/Prot_000.pdf